CLINICAL TRIAL: NCT06760455
Title: A Single-center, Double-blind, Placebo-controlled, Dose-escalation Phase I Clinical Study to Evaluate the Safety and Tolerability of BPR-30221616 Injection in Healthy Subjects
Brief Title: A Safety and Tolerability Study of BPR-30221616 Injection in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Brilliant Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BPR-30221616-Ⅰ-001
Record Dates: First submitted 2024-12-19; First posted 2025-01-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BPR-30221616 Injection (Experimental)
  Interventions: Drug: BPR-30221616 Injection
- Sodium Chloride Injection (Placebo Comparator)
  Interventions: Drug: Sodium Chloride Injection

INTERVENTIONS:
Drug: BPR-30221616 Injection — BPR-30221616 will be administered by subcutaneous (SC) injection
  Arms: BPR-30221616 Injection
Drug: Sodium Chloride Injection — Sodium Chloride Injection will be administered by SC injection
  Arms: Sodium Chloride Injection

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics、 pharmacodynamics and immunogenicity of BPR-30221616 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy subjects.
* Age 18 to 65 years.
* Male weight ≥ 50.0 kg ，female weight ≥ 45.0 kg ， BMI ≥18.0 and ≤30.0 kg/m^2.
* Females must be non-pregnant and non-lactating.
* Subjects must give informed consent prior to the trial and willing to give written informed consent form.
* Subjects who can communicate reliably with the investigator and comply with all study requirements .

Exclusion Criteria:

* Subjects who have a clinically relevant history or presence of neurological,respiratory, gastrointestinal, cardiovascular, haematological, immunological, genitourinary,hepatic,renal, musculoskeletal diseases， or considered unfit for the study by the investigator with new disease within the 7 days prior to dose administration.
* Subjects with a history of serious mental illness.
* Clinically-significant (CS) abnormalities in physical examination, vital signs, electrocardiogram, clinical laboratory examination , chest radiograph and abdominal ultrasound at screening visit.
* Alanine aminotransferase (ALT) >1.5× normal upper limit (ULN), or aspartate aminotransferase (AST) >1.5×ULN, or total bilirubin >1.5×ULN at screening visit.
* Glomerular filtration rate (eGFR) <90mL/min/1.73m2 at screening visit.
* Vitamin A level < lower limit of normal (LLN) at screening visit.
* Uncontrolled ventricular arrhythmias, or co-morbidities that may cause prolonged QT.
* Known history of allergic reactions to 2 or more drugs or to N-acetylated galactosamine (GalNAc) or oligonucleotides.
* Subjects who had undergone major surgery within 6 months prior to screening or planned to undergo surgery during the study period, and who had previously undergone surgery that would affect drug absorption, distribution, metabolism, or excretion (except surgery for appendicitis).
* Alcoholic or regular drinking within the 6 months of randomization; Or a positive baseline alcohol breath test.
* Subjects who have a history of drug abuse within the 12 months of screening or have a positive baseline drug screening result.
* Smoking >5 cigarettes a day.
* Known human immunodeficiency virus (HIV) ,Treponema pallidum Antibody (TP-Ab),hepatitis B surface antigen (HBsAg)or hepatitis C virus (HCV) infection at screening visit.
* Subjects who have donated 400 mL or more of blood within the 3 months prior to dose administration or plan to donate until 6 months after dose administration.
* From the signing of informed consent, throughout the study until 12 months after dose administration , unwilling to use appropriate and effective contraceptions.
* Received an investigational agent or device intervention within 3 months of screening.
* Received prescription drugs within 4 weeks of randomization.
* Received over-the-counter drugs(unless deemed not clinically relevant by the investigator) within 7 days of randomization.
* Received any oligonucleotides[including small interfering ribonucleic acid(siRNA) and antisense oligonucleotides].
* Intolerance to subcutaneous injection.
* Had a special diet (such as grapefruit and products containing grapefruit, chocolate, any food containing caffeine or rich in xanthines (such as animal liver)) or had strenuous activity within 48 hours prior to dose administration , or with other factors affecting drug absorption, distribution, metabolism, excretion.
* Any physical or mental illness or condition that, as determined by the study physician, is likely to increase the risk of the study, interfere with the subject's adherence to the protocol, or interfere with the subject's completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-01-24 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Participants With Adverse Events (AE) | Up to Day 360
Incidence of Participants With Serious Adverse Events (SAE) | Up to Day 360
Incidence of Participants With Clinically Significant laboratory tests, electrocardiogram (ECG), physical examination, vital signs | Up to Day 360

SECONDARY OUTCOMES:
Maximum plasma concentration （Cmax）of BPR-30221616 | Day 1 through to Day 3
Time to maximum plasma concentration（Tmax） of BPR-30221616 | Day 1 through to Day 3
Area under the plasma concentration-time curve（AUC）of BPR-30221616 | Day 1 through to Day 3
Elimination rate constant (λz) of BPR-30221616 | Day 1 through to Day 3
Elimination half-life (t1/2) of BPR-30221616 | Day 1 through to Day 3
Apparent volume of distribution during terminal phase (Vz/F) of BPR-30221616 | Day 1 through to Day 3
Clearance (CL/F) of BPR-30221616 | Day 1 through to Day 3
Mean residence time from zero to infinity (MRT0-∞) of BPR-30221616 | Day 1 through to Day 3
Cumulative amount of the dose excreted unchanged in urine (Ae) of BPR-30221616 | Day 1 through to Day 3
Cumulative fraction of the dose excreted unchanged in urine (Fe) of BPR-30221616 | Day 1 through to Day 3
Renal clearance(CLr) of BPR-30221616 | Day 1 through to Day 3
Effect of BPR-30221616 on serum transthyretin（TTR） levels as measured by reduction from baseline in serum TTR | Day 1 through to Day 540
Number of participants who develop serum anti-BPR-30221616 antibodies | Day 1 through to Day 360

OTHER OUTCOMES:
Effect of BPR-30221616 on serum Vitamin A levels as measured by reduction from baseline in serum Vitamin A | Day 1 through to Day 540
Effect of BPR-30221616 on serum Retinol-Binding Protein（RBP） levels as measured by reduction from baseline in serum RBP | Day 1 through to Day 540

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided